CLINICAL TRIAL: NCT02603822
Title: Performance of 13C Mannitol for in Vivo Measurement of Small Intestinal Permeability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Madhusudan (Madhu) Grover, MBBS, Madhusudan Grover, MBBS, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-003603
Record Dates: First submitted 2015-09-22; First posted 2015-11-13 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Impaired Small Intestinal Permeability
MeSH Terms: interventions — Indomethacin; Lactulose

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteers (Experimental): Subjects will receive a saccharide solution of 12C mannitol 100 mg, 13C mannitol 100 mg, and lactulose 1 g in 250ml of water at visits 2, 5, and 7 prior to permeability testing. The subjects will also receive Indomethacin capsules prior to visit 5.
  Interventions: Dietary Supplement: 12C mannitol; Drug: Indomethacin; Dietary Supplement: 13C mannitol; Dietary Supplement: Lactulose

INTERVENTIONS:
Dietary Supplement: 12C mannitol — 12C mannitol 100 mg
Drug: Indomethacin — Subjects will receive six 25 mg capsules of Indomethacin (immediate release). The subjects will take 3 capsules 8 hours before the timing of visit 5 (before fasting), and 3 additional capsules 30 minutes before visit 5.
  Other Names: Indocin
Dietary Supplement: 13C mannitol — 13C mannitol 100 mg
Dietary Supplement: Lactulose — lactulose 1 g

SUMMARY:
The investigators' overall objective with this study is to determine performance characteristics of small intestine permeability measurement using 13C mannitol and 12C (regular) mannitol.

DETAILED DESCRIPTION:
An impaired intestinal permeability is implicated in the pathophysiology of a number of disorders such as celiac disease, environmental enteropathy, inflammatory bowel disease, obesity, and HIV. Current measurements of intestinal permeability rely on urinary excretion of naturally available, orally ingested, non-absorbable sugars (e.g. lactulose, mannitol). However, dietary intake of these sugars limits interpretation from these assays.

Subjects will have an esophagogastroduodenoscopy (EGD) with biopsies and provide a baseline urine sample. They will be asked to ingest 3 saccharides (12C mannitol 100 mg,13C mannitol 100 mg and lactulose 1 g) in 250 ml of water. Urine samples will be obtained every 30 min. in the Clinical Research and Trials Unit (CRTU) for 0-2 hours. Subjects will collect 2-8 hour sample in provided container. Another container will be provided to collect the 8-24 hour urine which will be returned the following morning. Subjects will undergo an Indomethacin challenge intervention. They will be instructed to take three 25 mg capsules 8 hours before their next visit (just before fasting). They will take 3 additional 25 mg capsules 30 min. before the repeat in vivo permeability testing. Repeat EGD with duodenal biopsies will be done. Long term follow-up will be done within 4-6 weeks of previous testing, where subjects will once again be asked to complete the in vivo permeability testing.

ELIGIBILITY:
Healthy Volunteers

Inclusion criteria:

* Age (yr) 18 to 65
* No abdominal surgery (except appendectomy and cholecystectomy, others may be considered)

Exclusion criteria:

* History of irritable bowel syndrome (IBS), inflammatory bowel disease (IBD) (Crohn's disease or ulcerative colitis), microscopic colitis or celiac disease.
* Use of tobacco products within the past 6 months (since nicotine may affect intestinal permeability)
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) or aspirin within seven days of first permeability test (as NSAIDs affect intestinal permeability) and second permeability test (except those administered for the study)
* Use of oral corticosteroids within the previous 6 weeks
* Ingestion of artificial sweeteners such as Splenda® (sucralose), NutraSweet® (aspartame), lactulose or mannitol within two (2) days of each permeability test and endoscopy procedure date, e.g., foods to be avoided are sugarless gums or mints and diet soda
* Ingestion of any prescription, over the counter, or herbal medications which can affect gastrointestinal transit within 7 days each permeability test and endoscopy procedure date. This includes drugs such as serotonin (5-HT) agents, narcotics, anticholinergics, anti-nausea medications, any medications for diarrhea or constipation.
* Antibiotics within 7 days each permeability test and endoscopy procedure date
* Bleeding disorders or medications that increase risk of bleeding from mucosal biopsies.
* Score > 8 for anxiety or depression on Hospital Anxiety and Depression scale.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08; Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Small intestine permeability as measured by change in cumulative excretion of mannitol 0-2 hours | baseline, approximately 2 hours

SECONDARY OUTCOMES:
Colonic permeability as measured by change in mannitol excretion between 8 and 24 hours | 8 hours, approximately 24 hours
Change in mannitol excretion at 24 hours | baseline, approximately 24 hours
Change in lactulose-mannitol excretion assay at 2 hours | baseline, approximately 2 hours
  The ratio of urinary excretion of lactulose to mannitol was used to measure intestinal mucosal permeability, with higher ratios indicative of increased intestinal permeability.
Change in hour lactulose-mannitol excretion assay between 8 and 24 hours | 8 hours, approximately 24 hours
  The ratio of urinary excretion of lactulose to mannitol was used to measure intestinal mucosal permeability, with higher ratios indicative of increased intestinal permeability.

CONTACTS AND LOCATIONS:
Overall Officials: Madhusudan Grover, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided